CLINICAL TRIAL: NCT04770077
Title: Sniper Intubation for Training of Undergraduate Medical Student Randomized Controlled Trial
Brief Title: Sniper Intubation for Training of Undergraduate Medical Student
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, simon Halim Armanious, Lecturer, Ain Shams University
Other Study IDs: Sniper Intubation
Record Dates: First submitted 2021-02-23; First posted 2021-02-25 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Intubation;Difficult

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group S: Spray before intubation
  Interventions: Other: Intubation on manikin
- Group C: Intubation directly
  Interventions: Other: Intubation on manikin

INTERVENTIONS:
Other: Intubation on manikin — Training of medical student to focus on manikin vocal cord before intubation
  Other Names: Simulator

SUMMARY:
Students trained to focus on vocal cord before intubation

DETAILED DESCRIPTION:
Student trained to spray vocal cords with 3 ml normal saline over 30 seconds before intubation then allow them to introduce endotracheal tube

ELIGIBILITY:
Inclusion Criteria:

* medical student

Exclusion Criteria:

* previous training on endotracheal intubation

Ages: 18 Years to 25 Years | Sex: All
Age Groups: Adult
Study Population: Undergraduate medical student
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Rate of successful intubation | Less than 120 seconds

SECONDARY OUTCOMES:
Number of attempts | 120 seconds
Time to intubation | 120 seconds

IPD SHARING:
Plan to Share IPD: Undecided
Either through email contact with the corresponding author or through online Data sharing site {www.synapse.com}